CLINICAL TRIAL: NCT02792712
Title: Ticagrelor Versus Clopidogrel in Myocardial Salvage in Patients With ST-elevation Myocardial Infarction (STEMI) Undergoing Primary Percutaneous Coronary Intervention: A Magnetic Resonance Imaging Study (TIGER Study)
Brief Title: Ticagrelor Versus Clopidogrel in Myocardial Salvage in Patients With STEMI Undergoing Primary PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Tao-Cheng Wu, MD, PhD, Division of Cardiology, Department of Medicine, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2014-09-003A
Record Dates: First submitted 2016-05-18; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute myocardial infarction; Antiplatelet agents; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEMI_MRI_Ticagrelor (Experimental): A Magnetic Resonance Imaging Study in myocardial salvage in patients with ST-Elevation myocardial infarction (STEMI) undergoing pRimary percutaneous coronary intervention - Ticagrelor Arm
  Interventions: Drug: Ticagrelor
- STEMI_MRI_Clopidogrel (Active Comparator): A Magnetic Resonance Imaging Study in myocardial salvage in patients with ST-Elevation myocardial infarction (STEMI) undergoing pRimary percutaneous coronary intervention - Clopidogrel Arm
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 180 mg LD，then 90 mg BID
  Arms: STEMI_MRI_Ticagrelor
Drug: Clopidogrel — Clopidogrel 300 mg LD，then 75 mg QD
  Arms: STEMI_MRI_Clopidogrel

SUMMARY:
Therefore, in this study, we try to evaluate the impact of clopidogrel loading dose 300mg vs. ticagrelor 180 mg on myocardial injury as measured by contrast-enhanced magnetic resonance imaging (CE-MRI) in STEMI patients undergoing primary PCI.

DETAILED DESCRIPTION:
All STEMI patients will be loaded with dual oral antiplatelet therapy of 300 mg aspirin combined with either 300 mg clopidogrel or 180 mg ticagrelor before PCI, followed by maintenance dose of 100 mg aspirin plus 75 mg clopidogrel QD or 90 mg ticagrelor BID. The duty interventional cardiologists will be responsible for patient randomization based on a pre-defined randomization chart. As it is a usual practice in Taiwan for door-to-balloon time to be within 90 minutes, we hence do not expect any impact on study results due to D2B time variation.

All STEMI patients will receive loading dose of dual oral antiplatelet therapy with 300 mg aspirin combined with either 300 mg clopidogrel or 180 mg ticagrelor before PCI, followed by maintenance dose of 100 mg aspirin plus 75 mg clopidogrel QD or 90 mg ticagrelor BID.

The primary variable is to compare myocardial salvage index (in %) as assessed by CE-MRI between 300-mg clopidogrel group and ticargrelor group. Enzymatic infarct size will also be assessed, and two methods will be used to decide that. The first is cardiac troponinI 72 hours after pain onset , while the other is peak CK level after pain onset. Sampling timing of CK will be judged by the caring physicians.

The secondary objectives include: myocardial infarct size (% of LV mass), the extent of MVO, the number of segments with >75% of infarct transmurality.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Adult patients aged 20 years or older
3. STEMI within 12 hours of onset, defined as:presence of chest pain for >30 minutes and <12 hours after symptom onset; ST-segment elevation >1 mm in ≥2 contiguous leads or presumably a new-onset left bundle-branch block on electrocardiogram.
4. STEMI patients planned for PPCI

Exclusion Criteria:

1. STEMI > 12 h of onset
2. History of renal dysfunction requiring dialysis
3. Evidence of malignant diseases
4. Unwillingness to give out consent
5. Contraindicated for ticagrelor or clopidogrel

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Compare myocardial infarct size (myocardial salvage index %) as assessed by CE-MRI between 300-mg clopidogrel group and 180-mg ticargrelor group | 4-10 days after the index event

CONTACTS AND LOCATIONS:
Locations (1):
- Teipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No